CLINICAL TRIAL: NCT01898052
Title: A Comparative Study on the Efficacy of Periarticular Single Anesthetic Drug Compared With Multimodal Drug Injection in Controlling Pain After Total Knee Arthroplasty: A Double Blinded Randomized Controlled Trial
Brief Title: The Efficacy of Periarticular Single Drug Compared With Multimodal Drug Injection in Controlling Pain After TKA
Acronym: TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, department of orthopeadic surgery, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: orthoTU03; orthoTU03 (Other: Tha)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Postoperative Pain
Keywords: pain control; periarticular injection; Total knee arthroplasty; levobupivacaine; multimodal drug injection
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multimodal drug injection (Experimental): Multimodal drug injection Levobupivacaine 150 mg, epinephrine(1:1000) 0.6 mL(0.6 mg), morphine sulfate 5 mL(5 mg), ketorolac 1 mL (30 mg) and mixed with normal saline up to 100 mL
  Interventions: Drug: multimodal drug injection
- Single anaesthetic drug (Active Comparator): Single anaesthetic drug levobupivacaine 150 mg and epinephrine (1:1000) 0.6 ml (0.6 mg)
  Interventions: Drug: single anaesthetic drug

INTERVENTIONS:
Drug: single anaesthetic drug — inject periarticular tissue of the knee after implantation
  Other Names: levobupivacaine; chirocaine
  Arms: Single anaesthetic drug
Drug: multimodal drug injection — inject periarticular tissue of the knee
  Other Names: anaesthetic cocktail
  Arms: multimodal drug injection

SUMMARY:
The purpose of this study is to determine the periarticular multimodal drug injection has more efficacy for controlling pain after TKA than single anaesthetic drug injection.

DETAILED DESCRIPTION:
Many studies have to determine the efficacy of periarticular multimodal drug injection or single local anaesthetic drug comparing with placebo for pain controlled in TKA. But in this study would like to determine which one of both drugs are more efficacy.

In multimodal drug injection consist of levobupivacaine, morphine, ketorolac and epinephrine while single anaesthetic drug has levobupivacaine and epinephrine.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis of the knee who undergoing unilateral primary total knee arthroplasty
* age 50-85 years old

Exclusion Criteria:

* unable to perform spinal anaesthesia
* history of drug allergies; local anaesthesia, Non-steroidal anti-inflammatory drugs, morphine, epinephrine
* cognitive function impairment
* renal impairment (creatinine clearance < 30 mL/min)
* liver impairment, gastrointestinal bleeding

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
pain score | 48 hour after surgery
  pain score at rest and activity between 2 groups every 4 hours until 48 hours after surgery

SECONDARY OUTCOMES:
time to request analgesic drug | 48 hours
  time when patient request morphine from patient controlled analgesia after intra-operative drug injection

OTHER OUTCOMES:
drug consumption | 48 hours
  morphine consumption that record from patient controlled analgesia
knee score | 3 months
  Knee injury and osteoarthritis outcome score (KOOS) at pre-operation and post-operation 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Supakit Kanitnate, M.D., Principal Investigator — orthopaedics department
Locations (1):
- department of orthopaedic surgery, Faculty of medicine, Thammasat university, Khlong Luang, Changwat Pathum Thani, Thailand